CLINICAL TRIAL: NCT01130090
Title: Patient-ventilator Interactions in Long Term Non-invasive Ventilation (NIV): Influence of Back-up Frequency
Brief Title: Patient-ventilator Interactions in Long Term Non-invasive Ventilation: Influence of Back-up Frequency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ligue Pulmonaire Genevoise (Other)
Responsible Party: Jean-Paul Janssens / Professor, Division of Pulmonary Diseases; Geneva University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: CER- 08-131
Record Dates: First submitted 2010-05-03; First posted 2010-05-25 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Obesity; Non Invasive Ventilation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Adjustment of back-up respiratory rate on bi-level ventilator — 3 consecutive nights in randomized order, in either "S" (Spontaneous) mode, "ST" (Spontaneous/Timed) mode with a back-up rate under spontaneous respiratory rate of the patient, or in "ST" (Spontaneous/Timed) mode with a back-up rate at least 2 cycles/minute above spontaneous nocturnal respiratory rate. Each assessment will include complete polysomnographic recording (sleep study) as well as SpO2, PtcCO2, pneumotachograph (flow), mask pressure, quantitative assessment of patient-ventilator synchronisation, central or obstructive apnea and hypopnea, data of built-in software, and rating of patient comfort

SUMMARY:
In patients under bi-level pressure support ventilation for obesity hypoventilation syndrome, this study aims to determine if it is better, in terms of efficacy and patient-ventilator synchronisation to use

* Spontaneous mode (S)
* Spontaneous/Timed mode (ST) with an intermediate back-up rate, slightly below the respiratory rate of the patient
* Timed mode (T), with a ventilator respiratory rate above that of the patient. This issue has to our knowledge only been marginally studied without any consensus.

DETAILED DESCRIPTION:
Eligibility: patients under home bi-level pressure support ventilation for obesity hypoventilation in a stable clinical condition, aged over 18

Methods:

Three consecutive sleep studies in a randomised sequence with usual parameters Inspiratory Positive Airway Pressure(IPAP), Expiratory Positive Airway Pressure (EPAP) and change of only back up respiratory rate (RR): one night in a spontaneous mode, one with an intermediate RR, and one with a RR above that of the patient

Endpoints:

Quality of sleep and sleep structure (polysomnography), patient-ventilator synchronisation and respiratory events under NIV, efficacy of ventilation: oxygen saturation measured by pulse oxymetry (SaO2); transcutaneous capnography (PtcCO2), and comfort.

ELIGIBILITY:
Inclusion Criteria:

* Obesity-hypoventilation (OHS) patients, in stable clinical condition, treated with domiciliary nocturnal non invasive ventilation for at least two months

Exclusion Criteria:

* OHS patients: unstable cardio-respiratory status and/or acute cardio-respiratory failure three months before inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Sleep structure | Night 1
  Quantification of quality of sleep assessed by polysomnography (sleep stages, arousals)
Sleep structure | Night 2
  Quantification of quality of sleep assessed by polysomnography (sleep stages, arousals)
Sleep structure | Night 3
  Quantification of quality of sleep assessed by polysomnography (sleep stages, arousals)

SECONDARY OUTCOMES:
Transcutaneous capnography (PtcCO2) | Night 1
  Mean PtcCO2 during Night 1
Transcutaneous capnography (PtcCO2) | Night 2
  Mean PtcCO2 during night 2
Transcutaneous capnography (PtcCO2) | Night 3
  Mean PtcCO2 during night 3
Correlation between microarousal index and autonomic arousal index | Night 1
  Correlation between microarousal index (assessed by EEG) and autonomic arousal index under NIV (assessed by pulse plethysmography)
Correlation between microarousal index and autonomic arousal index | Night 2
  Correlation between microarousal index (measured by EEG) and autonomic arousal index (measured by pulse plethysmography)
Correlation between microarousal index and autonomic arousal index | Night 3
  Correlation between microarousal index (measured by EEG) and autonomic arousal index (measured by pulse plethysmography)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Janssens, MD, Study Director — University Hospital, Geneva
Locations (1):
- Geneva University hospital - Sleep laboratory, Geneva, Switzerland

REFERENCES:
- [Derived] Georges M, Adler D, Contal O, Espa F, Perrig S, Pepin JL, Janssens JP. Reliability of Apnea-Hypopnea Index Measured by a Home Bi-Level Pressure Support Ventilator Versus a Polysomnographic Assessment. Respir Care. 2015 Jul;60(7):1051-6. doi: 10.4187/respcare.03633. Epub 2015 Mar 3. PMID 25737571
- [Derived] Contal O, Adler D, Borel JC, Espa F, Perrig S, Rodenstein D, Pepin JL, Janssens JP. Impact of different backup respiratory rates on the efficacy of noninvasive positive pressure ventilation in obesity hypoventilation syndrome: a randomized trial. Chest. 2013 Jan;143(1):37-46. doi: 10.1378/chest.11-2848. PMID 22556317